CLINICAL TRIAL: NCT06249633
Title: A Pilot Study of Inhaled Nitric Oxide for ARDS-related Pulmonary Hypertension
Brief Title: Inhaled Nitric Oxide for ARDS-related Pulmonary Hypertension
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yuri Matusov (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor-Investigator, Yuri Matusov, Principal Investigator, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001807
Record Dates: First submitted 2024-01-12; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-01

CONDITIONS: Acute Respiratory Distress Syndrome; Pulmonary Hypertension
MeSH Terms: conditions — Respiratory Distress Syndrome; Hypertension, Pulmonary | interventions — Nitric Oxide; Endothelium-Dependent Relaxing Factors

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- iNOMAX (Experimental)
  Interventions: Drug: Nitric Oxide

INTERVENTIONS:
Drug: Nitric Oxide — Inhaled nitric oxide
  Other Names: iNOMAX

SUMMARY:
Open-label pilot study of early inhaled nitric oxide (iNO) for patients developing de novo pulmonary hypertension during Acute Respiratory Distress Syndrome (ARDS.) The study aims to determine whether iNO has possible hemodynamic and clinical benefits when given early in the course of ARDS to patients with evidence of elevated pulmonary artery pressure.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ARDS based on the Berlin criteria
* Mechanically ventilated
* Age ≥ 18 years

Exclusion Criteria:

* Primary cardiogenic shock
* History of more than mild pulmonary hypertension preceding ARDS diagnosis
* Presence of pre-existing significant valvular disease
* Presence of pre-existing left ventricular dysfunction or significant hypertrophy
* Consent cannot be obtained from the patient or his/her surrogates
* Refusal of consent
* Opinion of treating physicians that enrolling the patient in the study would be detrimental to his/her outcome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Determining improvement in pulmonary artery pressure in response to iNO | Approximately 4 days
  Pulmonary artery systolic pressure (in mmHg) will be determined by repeat echocardiography after initiation of iNO.
Determining improvement in tricuspid annular plane systolic excursion in response to iNO | Approximately 4 days
  Changes in tricuspid annular plane systolic excursion (in cm) will be determined by repeat echocardiography after initiation of iNO.
Determining improvement in right ventricular fractional area change in response to iNO | Approximately 4 days
  Changes in right ventricular fractional area change (in %) will be determined by repeat echocardiography after initiation of iNO.

SECONDARY OUTCOMES:
Improvement in urine output in response to iNO | Approximately 4 days
  Urine output changes will be determined by continuous bedside evaluation of urine output (in ml/hr) before and after initiation of iNO.
Improvement in serum creatinine in response to iNO | Approximately 4 days
  Changes in serum creatinine (in mg/dL) will be determined by laboratory analysis following initiation of iNO.

CONTACTS AND LOCATIONS:
Overall Officials: Yuri Matusov, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States